CLINICAL TRIAL: NCT04556721
Title: Assessing the Post-Surgical Trend of Sugammadex Concentration in Dialysis Dependent Patients
Brief Title: A Pharmacokinetic Study of Sugammadex in Dialysis Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty and lack of recruitment of the patients
Sponsor: Tetsuro Sakai (Other)
Responsible Party: Sponsor-Investigator, Tetsuro Sakai, Professor, Anesthesiology and Perioperative Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19090331
Record Dates: First submitted 2020-07-22; First posted 2020-09-21 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Renal Disease
Keywords: Sugammadex; Bridion; hemodialysis; renal disease; rocuronium; Sugammadex-Rocuronium complex
MeSH Terms: conditions — Kidney Diseases | interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sugammadex (Experimental): After surgery and general anesthesia, a clinically-appropriate dose of Sugammadex will be utilized to reverse the rocuronium neuromuscular blockade. Either 2 mg/kg or 4 mg/kg dosing will be used based on the level of neuromuscular blockade at the time of reversal. Administer as single IV bolus injection infused over 10 seconds into existing IV line. Dose is based on actual body weight (mg/kg).
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — On the day of surgery, after the establishment of general anesthesia, patients will be paralyzed via rocuronium. At the cessation of the case, an appropriate dose of Sugammadex will be utilized to reverse the rocuronium neuromuscular blockade.
  Other Names: Bridion

SUMMARY:
The primary objective of this prospective study is to assess the trend of sugammadex (and its complex with rocuronium) concentration in surgical patients with routine outpatient hemodialysis. Patients with end stage renal disease who are to receive general anesthesia and muscle paralysis will have their paralysis by rocuronium reversed with sugammadex. Patients will then have blood drawn during their next three routine hemodialysis sessions to assess for the plasma concentration of sugammadex or the sugammadex-rocuronium complex over time.

DETAILED DESCRIPTION:
Patients with end-stage renal disease often have several additional comorbidities and stand to benefit immensely from this established superior drug. Prior studies have not been able to correlate negative adverse events with sugammadex in patients with end-stage renal disease. More work needs to be done, however, to assess the fate of this renally excreted molecule. It has been shown that there is potential to clear sugammadex with high flux dialysis. We hypothesize that post-surgical patients with end-stage renal disease will see a significant decrease in plasma sugammadex concentration after routine outpatient dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Currently on hemodialysis renal replacement therapy
* To be undergoing a surgical procedure with the intent of starting hemodialysis postoperatively
* To be undergoing a surgical procedure requiring general anesthesia
* To have neuromuscular blockade for the surgical procedure

Exclusion Criteria:

* Diagnosed with a blood-borne infection (Hepatitis B or C, HIV)
* Allergy to rocuronium or sugammadex
* Planned renal transplant procedure
* Peritoneal dialysis patient
* Starting hemoglobin value of less than 8.0 g/dl
* Women who are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Plasma sugammadex concentration change from day of surgery to postoperative day 1 or 2 dialysis session | Day of surgery and postoperative day 1 or 2 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).
Plasma sugammadex concentration change from postoperative day 1 or 2 dialysis to postoperative day 3 or 4 dialysis session | Postoperative day 1 or 2 dialysis session and postoperative day 3 or 4 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).
Plasma sugammadex concentration change from postoperative day 3 or 4 dialysis session and postoperative day 5 or 6 dialysis session | Postoperative day 3 or 4 dialysis session and postoperative day 5 or 6 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).
Plasma sugammadex-rocuronium complex concentration change from day of surgery and postoperative day 1 or 2 dialysis session | Day of surgery and postoperative day 1 or 2 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).
Plasma sugammadex-rocuronium complex concentration change from postoperative day 1 or 2 dialysis to postoperative day 3 or 4 dialysis session | Postoperative day 1 or 2 dialysis session and postoperative day 3 or 4 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).
Plasma sugammadex-rocuronium complex concentration change from postoperative day 3 or 4 dialysis session and postoperative day 5 or 6 dialysis session | Postoperative day 3 or 4 dialysis session and postoperative day 5 or 6 dialysis session
  Plasma samples will be analyzed for concentrations of metabolites in units of microgram/milliliters (mcg/mL).

SECONDARY OUTCOMES:
Number of participants experiencing any number of AEs deemed related to sugammadex drug | Day of surgery through up to post-operative day 10
  Adverse events will be reviewed in the subject electronic medical records (EMR) and relation to the study drug will be determined by the investigator and recorded by research staff. Any untoward medical occurrence resulting from the study drug will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuro Sakai, MD, PhD, MHA, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No